CLINICAL TRIAL: NCT05704504
Title: Incorporating Ecological Momentary Assessment and Personalized Telephone Support Into Group-Based Exercise Intervention for Depressive Symptoms: A Pilot Randomized Controlled Trial
Brief Title: Incorporating Ecological Momentary Assessment and Personalized Telephone Support Into Group-Based Exercise Intervention for Depressive Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSY028
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Depression
Keywords: Depression; Exercise; Ecological momentary assessment; Randomised controlled trial
MeSH Terms: conditions — Depression; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-based exercise intervention with EMA and personalized telephone support (SUP) (Experimental): Participants in the SUP group will receive a 6-week group-based exercise intervention with ecological momentary assessment (EMA)and personalized telephone support.
  Interventions: Behavioral: Group-based exercise intervention with EMA and personalized telephone support (SUP)
- Group-based exercise intervention (EXE) (Active Comparator): Participants in the EXE group will receive a 6-week group-based exercise intervention.
  Interventions: Behavioral: Group-based exercise intervention (EXE)
- No intervention control group (CON) (No Intervention): Participants in the CON group will not be given any intervention during the study period but will be advised to remain their typical lifestyle throughout the trial period.

INTERVENTIONS:
Behavioral: Group-based exercise intervention with EMA and personalized telephone support (SUP) — Participants in the SUP group will receive a 6-week group-based exercise intervention with EMA and personalized telephone support. The intervention content includes three 120-minute group-based exercise training sessions delivered by a physical trainer and three 15-minute personalized telephone sessions delivered by research personnel. The first group exercise session will include (1) assessments of current physical fitness, (2) psychoeducation of depression, (3) education on the benefits of exercise on mental health, (4) demonstration and group low-intensity exercise training, and (5) smart goal setting. A booklet that summarizes the session content will be provided to participants. The second and third group exercise sessions will include (1) reviewing exercise goals and EMA data, (2) problem-solving barriers to exercise, (3) group discussion on exercise experience, (4) demonstration and group moderate-intensity exercise training, and (5) smart goal setting.
  Arms: Group-based exercise intervention with EMA and personalized telephone support (SUP)
Behavioral: Group-based exercise intervention (EXE) — Participants in the EXE group will receive a 6-week group-based exercise intervention. The intervention content includes three 120-minute group-based exercise training sessions delivered by a physical trainer at the Chinese University of Hong Kong. The first group exercise session will include (1) assessments of current physical fitness, (2) psychoeducation of depression, (3) education on the benefits of exercise on mental health, (4) demonstration and group low-intensity exercise training, and (5) smart goal setting. A booklet that summarizes the session content will be provided to participants. The second and the third group exercise sessions will include (1) reviewing exercise goals, (2) problem-solving barriers to exercise, (3) group discussion on exercise experience, (4) demonstration and group moderate-intensity exercise training, and (5) smart goal setting.
  Arms: Group-based exercise intervention (EXE)

SUMMARY:
The objective of this proposed pilot randomized controlled trial is to examine the efficacy and acceptability of using smartphone-delivered ecological momentary assessment (EMA) and personalized telephone support to promote adherence to a 6-week group-based exercise intervention for improving depressive symptoms.

Prior to all study procedures, eligible participants are required to complete an online informed consent via an in-house smartphone application, Longitudinax Pro. Around 60 eligible participants aged 18-65 years old with Patient Health Questionnaire (PHQ-9) total score ≥10 (Kroenke et al., 2001) and International Physical Activity Questionnaire (IPAQ) total score <600 MET/week (Lai et al., 2018; Macfarlane et al., 2007) will be randomly assigned to either 1) group-based exercise intervention with EMA and personalized telephone support (SUP), 2) group-based exercise intervention (EXE), or no intervention control group (CON) in a ratio of 1:1:1. The randomization will be performed by an independent assessor using a computer-generated list of numbers. The SUP and EXE groups will participate in a 6-week group-based exercise intervention. The intervention includes three biweekly group-based exercise sessions lasting for 120 minutes each (i.e., Week 1, 3, and 5). In addition, participants in the SUP will receive daily smartphone-delivered EMAs throughout the intervention period (i.e., 6-week) and 15-minute personalized telephone support delivered by a research personnel in Week 2, 4, and 6, respectively. Participants in the CON group will not be given any intervention during the study period but will be advised to remain their typical lifestyle throughout the trial period. The primary outcome of interest include depressive symptoms as measured by PHQ-9. The secondary outcomes will include anxiety symptoms, perceived insomnia severity, quality of life, functional impairment, and intervention evaluation at immediate post-intervention (Week 7) and 3-month follow-up assessments (Week 19).

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents
2. Aged ≥ 18 years
3. Able to read Chinese and type in Chinese or English
4. Have a Patient Health Questionnaire-9(PHQ-9) item score ≥10 indicating at least moderate level of depressive symptoms
5. Have an International Physical Activities Questionnaire- Chinese version (IPAQ-C) score <600 MET indicating physically inactive.
6. Have an Internet-enabled mobile device (iOS or Android operating system)
7. Willing to provide informed consent and comply with the trial protocol

Exclusion Criteria:

1. Received psychotherapy for depression in the past 6 months
2. A change in psychotropic drugs that target depression within 2 weeks before the baseline assessment
3. A PHQ-9 question 9 score higher than 2, indicating a moderate level of suicidal risk that requires active crisis management (referral information to professional mental health services will be provided)
4. Currently participating in another interventional study that may potentially improve mental health
5. Pregnancy
6. Self-disclosure of any psychiatric,medical or neurocognitive disorder(s) that makes participation unsuitable based on the team's clinical experience or interferes with adherence to the lifestyle modification (e.g., where exercise is not recommended by physicians)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, immediate post-intervention, and 3-month follow-up
  The PHQ-9, a 9-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Change in the Generalized Anxiety Disorder 7-item Scale (GAD-7) | Baseline, immediate post-intervention, and 3-month follow-up
  A brief 7-item instrument for screening for GAD and assessing its severity in clinical practice and research. Anxiety severity is categorized using scores of 5-9 (mild), 10-14 (moderate) and 15 or more (severe).
Change in the Insomnia Severity Index (ISI) | Baseline, immediate post-intervention, and 3-month follow-up
  ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in the Short Form (Six-Dimension) Health Survey - The Chinese (Hong Kong) Version | Baseline, immediate post-intervention, and 3-month follow-up
  A preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality. The SF-6D index, scored from 0.0 (worst health state) to 1.0 (best health state).
Change in the Short Multidimensional Inventory Lifestyle Evaluation (SMILE) | Baseline, immediate post-intervention, and 3-month follow-up
  The SMILE is a 43-item self-report questionnaire designed to measure 7 aspects of lifestyle, which included diet and nutrition (7-item), substance use (4-item), exercise (3-item), stress management (10-item), sleep management (5- item), social support (10-item), and environmental exposures (4-item). Each item is rated on a 4-point Likert scale. The possible response categories of each item are always (4), several days (3), seldom (2), and never (1).
Change in the Sheehan Disability Scale (SDS) | Baseline, immediate post-intervention, and 3-month follow-up
  SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life.
Change in the International Physical Activities Questionnaire - Chinese version (IPAQ-C) | Baseline, immediate post-intervention, and 3-month follow-up
  Participants' sitting time, walking time and moderate and vigorous physical activity are assessed by 5 questions from a short form of the International Physical Activity Questionnaire - Chinese version a short form of the IPAQ-C.
Change in the Treatment Acceptability and Adherence Scale (TAAS) | Baseline and immediate post-intervention
  TAAS is a self-reported, ten-item questionnaire that is rated by a seven-point Likert scale from 1 to 7, and it aims at evaluating the clients' attitude toward the treatment sessions by four domains, including acceptability, adherence, drop-out, and distress.
Change in Credibility-Expectancy Questionnaire (CEQ) | Baseline and immediate post-intervention
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success. Specific wording referencing "anxiety" was changed to refer to "depression".

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong